CLINICAL TRIAL: NCT05013112
Title: Ameliorating Metabolic Profiling After Kidney Transplantation (AMPKT): Protocol for an Open-label, Prospective, Randomized, 3-arm, Controlled Trial
Brief Title: Ameliorating Metabolic Profiling After Kidney Transplantation (AMPKT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Tao Lin, Professor Tao Lin, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WestChinaH-Metformin
Record Dates: First submitted 2021-07-20; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Kidney Transplantation; Metabolic Disorder; Metformin; Empagliflozin
MeSH Terms: conditions — Metabolic Diseases | interventions — Sodium-Glucose Transporter 2 Inhibitors; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo group (Placebo Comparator): Patients receive no additional therapy.
  Interventions: Other: Placebo
- Metformin group (Experimental): Patients receive metformin 500mg twice daily from discharge.
  Interventions: Drug: Metformin
- Empagliflozin (Experimental): Patients receive Empagliflozin once daily from discharge.
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — Empagliflozin 20mg once daily from discharge
  Arms: Empagliflozin
Drug: Metformin — Metformin 500mg twice daily from discharge
  Arms: Metformin group
Other: Placebo — Placebo group
  Arms: Placebo group

SUMMARY:
Advances in patient selection, organ procurement and preservation, surgical technique, immunosuppression, and infection prevention have conferred significant decrease in rejection, infection, and subsequently improve cause-specific graft failure rates after kidney transplantation (KT). However, cardiovascular diseases (CVD) remained the main burden impairing both short-and long-term survival. Compared with the general population, conventional CVD risk factors, including obesity, liver and muscle insulin resistance, dyslipidemia, hypertension, and diabetes mellitus, are all highly prevalent in this population. Risk factors of these metabolic disorders are generally reported, including common risk factors and those specifically for kidney transplants, including long-term exposure to steroids and calcineurin inhibitors.

Previous studies demonstrated that adenosine 5'-monophosphate (AMP)-activated protein kinase (AMPK) is a central regulator of multiple metabolic pathways and a key player in regulating cellular energy metabolism. Activation of AMPK by pharmacological agents may hold a considerable potential to reverse the metabolic abnormalities in chronic metabolic diseases. Metformin, a widely used antidiabetic drug, have been reported to act as an AMPK activator by inhibiting complex I of the mitochondrial electron transport chain in many tissues, including adipose, skeletal muscle, and heart. A recent small clinical trial observed that metformin administration did improve some of the metabolic profiles for glucocorticoid-treated patients with inflammatory disease but without pre-existing diabetes. In addition, another antidiabetic drug sodium-glucose-cotransporter-2 (SGLT-2) inhibitors can improve metabolic parameters and cardiovascular risk in patients with or without diabetes in preclinical and clinical studies. A small clinical trial reported that compared to metformin, significant improvement in anthropometric parameters and body composition, in overweight and obese women with polycystic ovary syndrome after 12 weeks of treatment with empagliflozin. Hence, metformin and SGLT2 agents may be used as potential adjuvant therapies to improve metabolic disorders after KT.

However, both metformin and SGLT-2 inhibitors were not recommended in patients with impaired kidney function considering their elimination and action mechanism. Although several preliminary clinical trials showed that metformin and SGLT-2 inhibitors can be used safely and improve glucose control after KT, but they are small-sample sized and only include patients with diabetes. We will conduct a prospective clinical trial with the first aim of exploring the safety of metformin and SGLT-2 inhibitors in kidney transplant recipients with or without diabetes, and the second aim of exploring their roles in improving metabolic profiling.

ELIGIBILITY:
Inclusion Criteria:

1. living-donor kidney transplantation;
2. eGFR level > 45ml/min/1.73m2 at discharge;
3. 18<Age<65 years;
4. receiving standard triad immunosuppressive regimen.

Exclusion Criteria:

1. previous therapy with metformin or SGLT 2 over the previous 3 months;
2. alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 or more of upper limit of normal;
3. Combined with HBV/HCV/HIV infection in the donor or recipient;
4. Malignancy history in the donor and recipient; 6) organ transplant history in the recipient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome was the differences in the visceral-to-subcutaneous fat area ratio over 12 months among three groups. | 12 months
  Based on previous study, visceral-to-subcutaneous fat area ratio, evaluated by CT, was generally reported as a surrogate for metabolic risk and was markedly raised in patients with long-term exposure to steroids. Hence, the primary outcome was the differences in the visceral-to-subcutaneous fat area ratio over 12 months among three groups.

SECONDARY OUTCOMES:
glycometabolic disorder | 12 months
  glycometabolic disorder was evaluated by fasting plasma glucose levels.
lipid metabolism | 12 months
  lipid metabolism was evaluated by serum triglyceride levels.
inflammatory status | 12 months
  inflammatory status was evaluated by C-reactive protein levels.